CLINICAL TRIAL: NCT03580096
Title: Effects of Core Stability Exercise in Patients With Parkinson's Disease
Brief Title: Core Stability and Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DF0074UG
Record Dates: First submitted 2018-06-15; First posted 2018-07-09 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Core Stability

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients were included in a core stability intervention. It will be done with different stages and increasing gradually.
  Interventions: Other: Core stability
- Control group (Active Comparator): Standard intervention consisting of exercises aimed at improving balance.
  Interventions: Other: Standard intervention

INTERVENTIONS:
Other: Core stability — Core stability intervention will be done with different stages and increasing gradually. The training program starts with exercises that isolate specific core muscles but progressing to include complex movements and incorporate core stability in dynamic tasks.
  Other Names: Core training
  Arms: Experimental group
Other: Standard intervention — Standard intervention will include active exercises based on active joint mobilizations, muscle stretching and motor coordination.
  Other Names: Conventional intervention
  Arms: Control group

SUMMARY:
Patients with Parkinson's Disease frequently present impaired postural control that leads to loss of stability and increased risk of falls.Core system, includes passive structures of the thoracolumbar spine and pelvis that work as a unit to stabilize the body and spine against forces generated from distal body segments as well as forces generated from expected or unexpected perturbations.The objective of this study was to evaluate the effects of an intervention based on core stability in patients with Parkinson's Disease.

DETAILED DESCRIPTION:
Core muscle coordination is important because lack of sufficient core muscle coordination can lead to decreased efficiency of postural control and functional activity. Clinical manifestations of patients with Parkinson's Disease include postural instability. Core system could be relevant to be included in an intervention. Thus, the objective of this study was to evaluate the effects of an intervention based on core stability in patients with Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease diagnosis.
* Stable medication usage
* Able to maintain standing independent

Exclusion Criteria:

* Cognitive impairment
* Comprehension deficits that prevented them from following verbal commands

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-07-08 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-11-04 (Actual)

PRIMARY OUTCOMES:
Change in dynamic balance | Change from baseline dynamic balance at 8 weeks
  Dynamic balance is going to be assessed with the Mini-Balance Evaluation System Test. It was developed to identify the postural control systems that underly poor functional balance. It contains four subscales: anticipatory postural control, reactive postural control, sensory orientation and stability in gait. It includes 14 items scored on a 3 level ordinal scale. The maximum total score is 28 points with higher scores indicating better balance.

SECONDARY OUTCOMES:
Balance confidence | Baseline, 8 weeks
  The perceived level of balance confidence is going to be assessed using the Activities-Specific Balance Confidence Scale (ABC). There are 16 items, representing daily activities. Participants are asked to answer, with a score from 0% (not confident at all) to 100% (completely confident) in increments of 10%. A score lower than 67% suggests substantial risk of falling.
Static balance | Baseline, 8 weeks
  Static balance is going to be assessed using the Wii Balance Board.The 4 sensors in the balance board can sense weight changes and show the distribution of body weight. It will be assessed standing balance with eyes opened and closed, and standing over a foam with eyes opened and closed. Higher time in a stable position indicates greater static balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, Granada, Spain

IPD SHARING:
Plan to Share IPD: No